CLINICAL TRIAL: NCT06196957
Title: Effect of Senobi Breathing Exercise Versus Buteyko Breathing Technique on the Functional Performance Among Chronic Obstructive Pulmonary Disease Patient.
Brief Title: Effect of Senobi Versus Buteyko Technique on Functional Performance of Chronic Obstructive Pulmonary Disease Patient.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ 0346 samar
Record Dates: First submitted 2023-11-22; First posted 2024-01-09 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Shortness of Breath
Keywords: Dyspnea, Quality of life, senobi,and buteyko
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko technique (Experimental): GROUP A'(Buteyko technique)
  Participant in group A will be instructed to perform the Buteyko breathing exercise.
  Patient either on the sitting position or standing position.
  Patient will be relaxed the shoulder and rest lower back against the back of chair.
  Close the mouth while only breathing through nose.
  Breath into the diaphragm and chest should be still.
  Exhale slowly, then hold the breath.
  Use the index finger and thumb to plug the nose, Hold the breath until there is urge to breath Then inhale
  Repeat several times. With in 15 minutes.
  Interventions: Combination Product: pursed lip breathing
- Senobi technique (Active Comparator): GROUP B (Senobi techniques)
  Senobi breathing exercise will be performed from standing, Arms will be extended firmly,
  The neck was extended so as face the ceiling. And the patient instructed to avoid over exertion
  Take a deep breath, hold for 3 second and then exhale through mouth.
  The time of exercise will be 15 minutes.
  Interventions: Combination Product: pursed lip breathing

INTERVENTIONS:
Combination Product: pursed lip breathing — pursed lip breathing
  Other Names: Senobi technique

SUMMARY:
Effect of Senobi breathing exercise versus Buteyko breathing technique on functional performance among chronic obstructive pulmonary patient.

DETAILED DESCRIPTION:
chronic obstructive pulmonary disease is a chronic inflammatory lung disease that cause obstructed airflow from the lungs. Symptoms include Breathing difficulty. cough, mucus production and wheezing. Its typically caused by long term exposure to irritating gasses or particulate matter, most often from cigarette smoker.

Emphysema and chronic bronchitis are two most common condition that contribute to chronic obstructive pulmonary disease. Chronic obstructive pulmonary disease is progressive disease that gets over a time. Clinical trials will be Conducted in Gulab Devi chest hospital in Lahore. Through the convenient sampling Technique. Which will be allocated through the random sampling two groups are involved group A and group B. In group A check the effect of Senobi techniques (stretch the body) and in group B check the effect of Buteyko technique. (Inhale the through the nose while mouth is closed) by using 6 mint walk test, Borg scale and quality of life questionnaire. Apply the technique to check the effectiveness of dyspnea and quality of life of patient The Buteyko technique offers a complementary method of reliving respiratory symptoms based on the voluntary control of breathing as well as considering the effect of environmental and dietary trigger. Data will be collected by the questionnaire and analyzed by using statistical package for the social science SPSS software version 21. The Buteyko method made its way to Australia to Europe and the unite states in 1990, it become best for the asthma and chronic obstructive pulmonary disease patient. The Senobi stretch exercise of the respiratory muscle improve the chest expansion and also improve the chest wall mobility in chronic obstructive pulmonary disease patient. Senobi breathing exercise was found to be effective for depression and it regulate the sympathetic nerve activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 -80
* COPD patient in stage 2 (GOLD criteria)
* Dyspnea (FEV1< 70 %)(26)
* Maximum expiratory pressure: 50%
* Smoker

Exclusion Criteria:

* Patient with Tumor
* Patient with Cardiac Arrhythmias Patient
* Patient with cancer
* insulin dependent diabetes
* patient with thyroid disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
CASA Q (cough and sputum ) | 4 weeks
  The cough and sputum assessment questionnaire (CASA-Q) was used to measure the severity and impact of cough and sputum in patients with COPD and chronic bronchitis. CASA-Q scores of each domain demonstrated significant association with HRQoL impairment CASA-Q was strongly lower when chronic bronchitis was present, but multivariate analyses demonstrated that the association of HRQoL impairment was greater with the cough impact domain score than with the usual definition of chronic bronchitis. The CASA-Q targets cough and sputum by an original approach assessing both the symptoms and impacts in dailyactivities within the last 7 days. Each item is answered ranging from never to always or from not at all to a lot / extremely as applicable each type is answered using five categories.
Dyspnea rating scale. | 4 weeks
  This scale is used for the measurement of the dyspnea ( shortness of breath ).This scale is questionnaire that consist of 5 breathlessness grade ,and the number 5 have maximum dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Sumera abdulhameed, ms, Principal Investigator — Riphah International University
Locations (1):
- Gulab devi chest hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cortopassi F, Gurung P, Pinto-Plata V. Chronic Obstructive Pulmonary Disease in Elderly Patients. Clin Geriatr Med. 2017 Nov;33(4):539-552. doi: 10.1016/j.cger.2017.06.006. Epub 2017 Aug 23. PMID 28991649
- [Background] Cowie RL, Conley DP, Underwood MF, Reader PG. A randomised controlled trial of the Buteyko technique as an adjunct to conventional management of asthma. Respir Med. 2008 May;102(5):726-32. doi: 10.1016/j.rmed.2007.12.012. Epub 2008 Jan 31. PMID 18249107
- [Background] Opat AJ, Cohen MM, Bailey MJ, Abramson MJ. A clinical trial of the Buteyko Breathing Technique in asthma as taught by a video. J Asthma. 2000;37(7):557-64. doi: 10.3109/02770900009090810. PMID 11059522